CLINICAL TRIAL: NCT02055534
Title: Nutritional Counseling in Systemic Immunoglobulin Light-chain (AL) Amyloidosis: a Prospective Randomized, Controlled Trial.
Brief Title: Nutritional Counseling in Systemic Immunoglobulin Light-chain Amyloidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVSMATT01 - amyloid nutr
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2014-02

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional counseling (Experimental): Nutritional counseling consists in: personalized dietary prescription associated with regular (every 3 weeks) dietetic advise by a registered dietician. Follow-up evaluations take place also during the visits scheduled by the Amyloidosis Center
  Interventions: Other: Nutritional counseling
- General dietary advices (Other): General dietary advices are provided. Follow-up evaluations take place during the visits scheduled by the Amyloidosis Center
  Interventions: Other: General dietary advices

INTERVENTIONS:
Other: Nutritional counseling — Nutritional counseling consists in: personalized dietary prescription associated with regular (every 3 weeks) dietetic advise by a registered dietician. Follow-up evaluations take place also during the visits scheduled by the oncologists
  Arms: Nutritional counseling
Other: General dietary advices — General dietary advices are provided. Follow-up evaluations take place during the visits scheduled by the oncologists
  Arms: General dietary advices

SUMMARY:
Poor nutritional status is common in patients with systemic immunoglobulin light-chain (AL) amyloidosis and has been associated with mortality and impaired quality of life (QoL). We investigated whether nutritional counseling is beneficial to the maintenance of nutritional status and QoL in AL outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve patients with with systemic immunoglobulin light-chain amyloidosis
* Availability to planned measurements and to written informed consent

Exclusion Criteria:

* Age < 18 years
* Indication to organ transplantation
* Indication to autologous stem cell transplantation
* Need to start or ongoing dialysis
* Ascites or massive edema
* Need to start or ongoing artificial nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 months
  Change in body weight at 12 months

SECONDARY OUTCOMES:
Quality of life | 12 months
  Change in quality of life at 12 months
Overall survival | 12 months
  Overall survival at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Italy; Giampaolo Merlini, MD, Study Chair — Amyloidosis Research and Treatment Center, Biotechnology Research Laboratories, Department of Molecular Medicine, Fondazione IRCCS Policlinico San Matteo and University of Pavia, Italy
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Caccialanza R, Palladini G, Klersy C, Cereda E, Bonardi C, Cameletti B, Quarleri L, Montagna E, Foli A, Milani P, Lavatelli F, Marena C, Merlini G. Malnutrition at diagnosis predicts mortality in patients with systemic immunoglobulin light-chain amyloidosis independently of cardiac stage and response to treatment. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):891-4. doi: 10.1177/0148607113501328. Epub 2013 Sep 26. PMID 24072737
- [Background] Caccialanza R, Palladini G, Klersy C, Cereda E, Bonardi C, Cameletti B, Montagna E, Russo P, Foli A, Milani P, Lavatelli F, Merlini G. Nutritional status independently affects quality of life of patients with systemic immunoglobulin light-chain (AL) amyloidosis. Ann Hematol. 2012 Mar;91(3):399-406. doi: 10.1007/s00277-011-1309-x. Epub 2011 Aug 9. PMID 21826471
- [Background] Caccialanza R, Palladini G, Klersy C, Cena H, Vagia C, Cameletti B, Russo P, Lavatelli F, Merlini G. Nutritional status of outpatients with systemic immunoglobulin light-chain amyloidosis 1. Am J Clin Nutr. 2006 Feb;83(2):350-4. doi: 10.1093/ajcn/83.2.350. PMID 16469994
- [Background] Sattianayagam PT, Lane T, Fox Z, Petrie A, Gibbs SD, Pinney JH, Risom SS, Rowczenio DM, Wechalekar AD, Lachmann HJ, Gilbertson JA, Hawkins PN, Gillmore JD. A prospective study of nutritional status in immunoglobulin light chain amyloidosis. Haematologica. 2013 Jan;98(1):136-40. doi: 10.3324/haematol.2012.070359. Epub 2012 Sep 14. PMID 22983575
- [Derived] Caccialanza R, Palladini G, Cereda E, Bonardi C, Milani P, Cameletti B, Quarleri L, Cappello S, Foli A, Lavatelli F, Klersy C, Merlini G. Nutritional counseling improves quality of life and preserves body weight in systemic immunoglobulin light-chain (AL) amyloidosis. Nutrition. 2015 Oct;31(10):1228-34. doi: 10.1016/j.nut.2015.04.011. Epub 2015 May 11. PMID 26250487